CLINICAL TRIAL: NCT02578888
Title: Early Palliative Medicine Intervention Using Idiographic Assessment for Women With High Risk Gynecologic Malignancies
Brief Title: Palliative Care in Improving Quality of Life in Patients With High Risk Primary or Recurrent Gynecologic Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nicole Nevadunsky, Principal Investigator, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-4421; NCI-2015-00729 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-4421 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2015-10-13; First posted 2015-10-19 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Cervical Carcinoma; Ovarian Carcinoma; Primary Peritoneal Carcinoma; Recurrent Cervical Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Uterine Corpus Carcinoma; Recurrent Vulvar Carcinoma; Uterine Corpus Cancer; Vulvar Carcinoma; Peritoneal Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms; Vulvar Neoplasms; Peritoneal Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palliative Therapy (Active Comparator): EORTCQLQ-30 and FAMCARE questionnaire every 6 weeks for 3 visits.
  Interventions: Other: Palliative Therapy; Other: Palliative Therapy + idiographic
- Palliative Therapy+ idiographic (Experimental): EORTC QLQ-30, and FAMCARE questionnaire every 6 weeks for 3 visits plus patients undergo idiographic assessment.
  Interventions: Other: Palliative Therapy; Other: Palliative Therapy + idiographic

INTERVENTIONS:
Other: Palliative Therapy — Palliative Therapy
  Other Names: Palliative Care; Symptom Management
Other: Palliative Therapy + idiographic — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized clinical trial studies a palliative care program in improving the quality of life of patients with high-risk gynecologic malignancies that is original or first tumor in the body (primary) or has come back (recurrent). Palliative care is care given to patients and their families facing the problems associated with life-threatening illness, through the prevention and relief of suffering by means of early identification and impeccable assessment and treatment of pain and other problems, physical, psychosocial and spiritual. Studying a palliative care program may help doctors learn more about patients quality of life, use of healthcare services, and the relief of pain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Validate a model of proactive palliative medicine referral. II. Quantify the impact of palliative care aggressive care at the end-of-life (PCARE) versus PCARE + idiographic assessment on quality of care and patient satisfaction.

III. Utilizing CMO data Investigators will create a cost model for patients randomized to PCARE versus patients refusing randomization.

IV. Determine the impact of a proactive model of palliative care consultation at the time of diagnosis on family/caregivers.

OUTLINE: Patients are randomized 1 of 2 arms.

GROUP I (usual PCARE): Patients complete European Organization for Research and Treatment of Cancer quality of life-30 (EORTCQLQ-30) and Family Satisfaction with Advanced Cancer Care (FAMCARE) questionnaire every 6 weeks for 3 visits.

GROUP II: (usual PCARE + idiographic assessment): Patients complete EORTC QLQ-30, and FAMCARE questionnaire as in Group I and undergo idiographic assessment. Beginning within 4 weeks of their visit with the gynecologic oncologist, patients are referred to outpatient palliative medicine consultation.

After completion of study, patients are followed up periodically .

ELIGIBILITY:
Inclusion Criteria:

* Women with of primary or recurrent diagnosis of ovarian, uterine, peritoneal, cervical or vulvar cancer with any of the following:

  * < 30 % projected 5 year survival based on histopathological stage
  * Non-pelvic recurrent malignancy
  * Persistent or progressive disease despite primary treatment with surgery, chemotherapy or
  * Palliative performance scale < 60
* Enrollment within 6 weeks of tumor board review

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Measure increased utilization (move from 18% to over 50%) of palliative medicine and increased proportion of patients receiving services more then 30 days before death as compared to historical controls. | Baseline
  To validate a model of proactive palliative medicine referral; We recorded that proactive referral will result in a clinically relevant increase of utilization of palliative medicine services (>70% of eligible women will have at least 1 consultation) and facilitate proxy assignment and improve pain/symptom control. There will be increased utilization of palliative care.
Measured by differential in aggresive care at end-of-life from direct hospital costs in the last 6 months of life between patients that are randomized and refuse randomization. | Up to 3 years
  We measured ACE and decreased direct hospital cost of care in the last 6 months of life between patients randomized and refusing randomization.
Evaluate costs related to procedures, laboratories, radiographic studies, intensive care admission, and blood transfusion to create a model of potential cost savings as generalized to patients with non-gynecologic cancers within the CMO. | Up to 3 years
  We utilized CMO data to create a cost model for patients randomized to PCARE versus patients refusing randomization. Costs related to potentially "preventable spends" will be obtained from the CMO database for eligible patients.
FAMCARE Survey will be administered, a 20 item scale measuring the degree to which family members are satisfied with the healthcare providers' behaviors. Comparison of family member scores between 2 arms, as well as at face value will be evaluated. | up to 3 years
  We administered a patient satisfaction scale

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Nevadunsky, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States